CLINICAL TRIAL: NCT00101348
Title: A Phase I, and Biologic Correlative Study of Erlotinib, in Combination With Cetuximab and Bevacizumab in Patients With Metastatic Renal Cell Carcinoma
Brief Title: Erlotinib and Cetuximab With or Without Bevacizumab in Treating Patients With Metastatic or Unresectable Kidney, Colorectal, Head and Neck, Pancreatic, or Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02639; NCI-2012-02639 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000401514; NCI-6588; CTRC-IDD-0332 (Other: Cancer Therapy and Research Center at The UT Health Science Center at San Antonio); 6588 (Other: CTEP); U01CA069853 (NIH); P30CA054174 (NIH)
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2012-12

CONDITIONS: Metastatic Squamous Neck Cancer With Occult Primary Squamous Cell Carcinoma; Recurrent Adenoid Cystic Carcinoma of the Oral Cavity; Recurrent Basal Cell Carcinoma of the Lip; Recurrent Colon Cancer; Recurrent Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Recurrent Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Recurrent Lymphoepithelioma of the Nasopharynx; Recurrent Lymphoepithelioma of the Oropharynx; Recurrent Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Recurrent Mucoepidermoid Carcinoma of the Oral Cavity; Recurrent Non-small Cell Lung Cancer; Recurrent Pancreatic Cancer; Recurrent Rectal Cancer; Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Stage III Adenoid Cystic Carcinoma of the Oral Cavity; Stage III Basal Cell Carcinoma of the Lip; Stage III Colon Cancer; Stage III Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Stage III Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Stage III Lymphoepithelioma of the Nasopharynx; Stage III Lymphoepithelioma of the Oropharynx; Stage III Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Stage III Mucoepidermoid Carcinoma of the Oral Cavity; Stage III Pancreatic Cancer; Stage III Rectal Cancer; Stage III Salivary Gland Cancer; Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Nasopharynx; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage III Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage III Verrucous Carcinoma of the Larynx; Stage III Verrucous Carcinoma of the Oral Cavity; Stage IIIB Non-small Cell Lung Cancer; Stage IV Adenoid Cystic Carcinoma of the Oral Cavity; Stage IV Basal Cell Carcinoma of the Lip; Stage IV Colon Cancer; Stage IV Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Stage IV Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Stage IV Lymphoepithelioma of the Nasopharynx; Stage IV Lymphoepithelioma of the Oropharynx; Stage IV Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Stage IV Mucoepidermoid Carcinoma of the Oral Cavity; Stage IV Non-small Cell Lung Cancer; Stage IV Pancreatic Cancer; Stage IV Rectal Cancer; Stage IV Renal Cell Cancer; Stage IV Salivary Gland Cancer; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Oropharynx; Stage IV Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IV Verrucous Carcinoma of the Larynx; Stage IV Verrucous Carcinoma of the Oral Cavity; Untreated Metastatic Squamous Neck Cancer With Occult Primary
MeSH Terms: conditions — Colonic Neoplasms; Esthesioneuroblastoma, Olfactory; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Rectal Neoplasms; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Renal Cell | interventions — Erlotinib Hydrochloride; Cetuximab; Bevacizumab

ARMS (1):
- Treatment (erlotinib hydrochloride, cetuximab, bevacizumab) (Experimental): Part 1: Patients receive oral erlotinib once daily on days 1-28. Patients also receive cetuximab IV over 3 hours on day 1 and over 1 hour on days 8, 15, and 22.
  Cohorts of 3-6 patients receive escalating doses of erlotinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  Part 2: Patients receive erlotinib as in part 1 at the MTD and cetuximab as in part 1. Patients also receive bevacizumab IV over 1½ hours on day 1 and over 1 hour on day 15.
  Cohorts of 3-6 patients receive escalating doses of bevacizumab until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  In both groups, courses repeat every 28 days in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: erlotinib hydrochloride; Biological: cetuximab; Biological: bevacizumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given orally
  Other Names: CP-358,774; erlotinib; OSI-774
Biological: cetuximab — Given IV
  Other Names: C225; C225 monoclonal antibody; IMC-C225; MOAB C225; monoclonal antibody C225
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase I/II trial studies the side effects, best way to give, and best dose of erlotinib and bevacizumab when given with cetuximab and how well giving erlotinib and cetuximab together with or without bevacizumab works in treating patients with metastatic or unresectable kidney, colorectal, head and neck, pancreatic, or non-small cell lung cancer. Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as cetuximab and bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Cetuximab and bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving erlotinib together with cetuximab and/or bevacizumab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of erlotinib when combined with cetuximab in patients with metastatic or unresectable renal cell, colorectal, head and neck, pancreatic, or non-small cell lung cancer (part 1).

II. Determine the MTD of bevacizumab when combined with cetuximab and erlotinib in these patients (part 2).

III. Determine the toxic effects, both quantitatively and qualitatively, of these regimens in these patients.

IV. Determine the antitumor activity of these regimens, in terms of tumor response, short-term survival, and progression-free survival, in these patients.

SECONDARY OBJECTIVES:

I. Compare, preliminarily, the toxicity and antitumor activity profiles of these regimens in these patients.

OUTLINE: This is an open-label, multicenter, dose-escalation study of erlotinib and bevacizumab.

Part 1: Patients receive oral erlotinib once daily on days 1-28. Patients also receive cetuximab IV over 3 hours on day 1 and over 1 hour on days 8, 15, and 22.

Cohorts of 3-6 patients receive escalating doses of erlotinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Part 2: Patients receive erlotinib as in part 1 at the MTD and cetuximab as in part 1. Patients also receive bevacizumab IV over 1½ hours on day 1 and over 1 hour on day 15.

Cohorts of 3-6 patients receive escalating doses of bevacizumab until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

In both groups, courses repeat every 28 days in the absence of unacceptable toxicity or disease progression.

After completion of study treatment, patients are followed at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* One of the following histologically confirmed diagnoses:

  * Renal cell cancer

    * Clear cell histology
    * Metastatic or unresectable disease AND meets 1 of the following criteria:

      * Recurrent disease
      * Refractory to interleukin-2 (IL-2)- or interferon-based therapy
      * Previously untreated AND not a candidate for IL-2-based therapy
  * Colorectal, head and neck, pancreatic, or non-small cell lung cancer

    * Metastatic or unresectable disease
    * Progression after prior standard treatment
* No evidence of CNS disease, including the following (part 2 only):

  * Primary brain tumor
  * Brain metastases
* Paraffin embedded tumor blocks available
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* More than 12 weeks
* Absolute neutrophil count ≥ 1,500 mm^3
* Platelet count ≥ 100,000 mm^3
* Bilirubin ≤ 1.5 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastasis is present)
* PTT and INR ≤ 1.5, unless receiving full-dose warfarin (part 2 only)
* Creatinine ≤ 1.5 times ULN
* Creatinine clearance ≥ 60 mL/min
* Calcium < 10 mg/dL (hypocalcemic agents allowed)
* No proteinuria*
* Protein < 1 g on 24-hour urine collection*
* No unstable angina pectoris
* No cardiac arrhythmia
* No symptomatic congestive heart failure
* None of the following are allowed for part 2:

  * Myocardial infarction within the past 6 months
  * New York Heart Association class II-IV heart disease
  * Serious cardiac arrhythmia requiring medication
  * Peripheral vascular disease ≥ grade II
  * Recent history of cerebrovascular accident
  * Uncontrolled hypertension (blood pressure ≥ 150/85 mm Hg despite medication)
  * Other clinically significant cardiovascular disease
* No gastrointestinal (GI) tract disease resulting in an inability to take oral medication
* No GI tract disease resulting in a requirement for IV alimentation
* No active peptic ulcer disease
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to study drugs
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies (part 2 only)
* No ongoing or active infection
* No active infection requiring parenteral antibiotics (part 2 only)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study treatment
* No significant traumatic injury within the past 28 days (part 2 only)
* No history of abnormalities of the cornea (e.g., dry eye syndrome, Sjögren's syndrome, or congenital abnormality [e.g., Fuch's dystrophy])
* No other malignancy within the past 3 years except nonmelanoma skin cancer or carcinoma in situ of the breast or cervix
* No psychiatric illness or social situation that would preclude study compliance
* No serious or non-healing wound ulcer or bone fracture (part 2 only)
* No other uncontrolled illness
* See Disease Characteristics
* More than 4 weeks since prior immunotherapy
* No prior cetuximab
* No prior bevacizumab
* Concurrent epoetin alfa or darbepoetin alfa allowed
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* More than 4 weeks since prior radiotherapy
* No prior surgical procedures affecting absorption
* Prior nephrectomy or resection of metastatic lesions allowed provided patient has fully recovered
* More than 7 days since prior core biopsy*
* More than 28 days since prior major surgery or open biopsy*
* No concurrent major surgery*
* Recovered from all prior therapy
* No prior erlotinib
* Concurrent bisphosphonates allowed
* Concurrent full-dose anticoagulants allowed provided the following criteria are met (part 2 only):

  * In-range INR (usually between 2 and 3) AND on a stable dose of warfarin or low molecular weight heparin
  * No active bleeding
  * No pathological conditions that carry a high risk of bleeding (e.g., tumor involving major vessels or varices)
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2005-01; Primary Completion 2007-10 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of erlotinib hydrochloride combined with cetuximab determined by dose-limiting toxicities (DLT) graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3 (Part I) | 28 days
  The occurrence and maximal grade of toxicity for the whole duration of treatment will be listed and tabulated by type.
MTD of bevacizumab combined with cetuximab and erlotinib hydrochloride determined by DLT graded according to the CTCAE version 3 (Part II) | 28 days
  The occurrence and maximal grade of toxicity for the whole duration of treatment will be listed and tabulated by type.

SECONDARY OUTCOMES:
Antitumor activity defined as the number and extent (complete or partial) objective responses as well as objective stable disease as measured by RECIST criteria | 6 months
  The estimated rate and their 95% confidence interval, will be reported.
Median time to progression | Up to 1 month
Progression-free survival | From the start of the treatment until the date the criteria for progression are met or the date the patient is taken off study for any reason, assessed up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Alain Mita, Principal Investigator — Cancer Therapy and Research Center at The UT Health Science Center at San Antonio
Locations (1):
- Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas, United States